CLINICAL TRIAL: NCT01097941
Title: Evaluation of the Effect of Age and Prior Immunity on the Response to Live or Inactivated A/California/07/09 H1N1 Influenza Vaccines in Children
Brief Title: Effect of Age and Prior Immunity on Response to H1N1 Vaccines in Children
Acronym: H1N1Children
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Live H1N1 vaccine expired and unable to get new supply
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, John Treanor, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URMC 09-007
Record Dates: First submitted 2010-03-30; First posted 2010-04-02 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: 2009 H1N1 Influenza
Keywords: Influenza; H1N1
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAIV/LAIV (Active Comparator)
  Interventions: Biological: Live Attenuated H1N1 Influenza Vaccine
- IIV/IIV (Active Comparator)
  Interventions: Biological: Influenza A (H1N1) 2009 Monovalent Vaccine
- IIV/LAIV (Active Comparator)
  Interventions: Biological: Influenza A (H1N1) 2009 Monovalent Vaccine/ Influenza A (H1N1) Monovalent Vaccine Live

INTERVENTIONS:
Biological: Live Attenuated H1N1 Influenza Vaccine — 0.2 ml dose of live monovalent vaccine delivered through nasal spray, 2 doses given 28 days apart
  Other Names: Influenza A (H1N1) 2009 Monovalent Vaccine Live, Intranasal
  Arms: LAIV/LAIV
Biological: Influenza A (H1N1) 2009 Monovalent Vaccine — 0.5 ml IM, 2 doses given 28 days apart
  Other Names: Influenza vaccine
  Arms: IIV/IIV
Biological: Influenza A (H1N1) 2009 Monovalent Vaccine/ Influenza A (H1N1) Monovalent Vaccine Live — 0.5 ml IM given X1 with 0.1 ml intranasally given 28 days later
  Other Names: Influenza Vaccine
  Arms: IIV/LAIV

SUMMARY:
A total of 51 children between the ages of 4 and 9 will be randomized to receive a two dose schedule of either licensed live attenuated A/California/07/09 influenza vaccine (LAIV) or licensed inactivated A/California/07/09 influenza vaccine (IIV) or IIV followed by LAIV separated by 28 days. Children with prior vaccination or natural infection with novel H1N1 influenza will be excluded. Randomization will be stratified by pre-existing HAI titers to the previous winter's seasonal H1N1 A/Brisbane/57/07 reference virus.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, prospective, open-label evaluation of the clinical tolerability, vaccine virus shedding, and serum and mucosal antibody response to vaccination with either live monovalent novel H1N1 influenza vaccine (LAIV) or monovalent inactivated novel H1N1 influenza vaccine (IIV) in healthy children between the ages of 4 and 9 years. Children will be screened for antibody to A/Brisbane/57/07 (H1N1) and A/California/07/09 (H1N1) prior to randomization. Children with evidence of prior exposure to the 2009 pandemic H1N1 virus will be excluded. Those with antibodies to A/Brisbane/57/07 (H1N1) will be stratified by preexisting antibody. Vaccine will be administered on days 0 and 28.

Safety of vaccination will be assessed using symptoms collected by parents for 7 days after each dose of vaccine. Serum will be obtained prior to and on day 28 following each dose of vaccine and assessed for antibody by HAI, ELISA, B-cell ELISPOT and neutralization techniques. Nasal secretions will be obtained by nasal aspiration prior to and on day 28 after each dose and assessed for HA-specific IgA antibody by ELISA. Nasal swabs will be obtained on days 2, 4, and 7 after each dose of live vaccine and assessed for the presence and magnitude of vaccine virus shedding of the live attenuated vaccine by rtRT-PCR and TCID50 on MDCK cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 9 years, inclusive.
* Pre-vaccination serum HAI titer to A/California/07/09 of 8 or less
* No prior history of laboratory documented infection with novel H1N1 virus or immunization with novel H1N1 vaccine.
* in good health, as determined by: vital signs (heart rate <140 bpm; blood pressure: systolic ≥ 90 mm Hg and ≤140 mm Hg; diastolic ≤ 90 mm Hg; oral temperature <100.0ºF); medical history; and targeted physical examination, when necessary, based on medical history. Stable medical condition is defined as: no recent increase in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months.
* subject/parents are able to understand and comply with the planned study procedures, including being available for all study visits.
* subject/parents have provided informed consent prior to any study procedures. (An assent will be obtained for all children 6 years and older)

Exclusion Criteria:

* a previous history of vaccination against novel H1N1 virus or a laboratory documented history of previous novel H1N1 infection.
* History of egg allergy or allergy to other components of vaccine.
* History of wheezing.
* immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy.
* has an active neoplastic disease.
* has long-term (greater than 2 weeks) use of oral or parenteral steroids, or high-dose inhaled steroids (>800 mg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* received immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
* has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days (or 56 days for vaccine naïve recipients).
* has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include chronic conditions recognized as risk factors for influenza complications or as contraindications for live vaccination, including chronic cardiac (exclusive of hypertension) or pulmonary conditions (including asthma), diabetes mellitus, or renal impairment.
* has an acute illness or an oral temperature greater than 99.9 degrees F (37.7 degrees C) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated symptoms resolved are eligible to enroll as long as treatment is completed and symptoms resolve > 3 days prior to enrollment.
* is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period.
* has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* has a previous history of Guillain-Barré syndrome within 6 weeks of receipt of influenza vaccination.
* has any condition that the principal investigator (PI) believes may interfere with successful completion of the study.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for assessment of the live attenuated vaccine take will be the AUC of the live vaccine virus shedding determined by 50% tissue culture infectious dose (TCID ) on MDCK cells at 33 degrees C | nasal swabs obtained at days 2 post vaccination
The primary endpoint for assessment of the live attenuated vaccine take will be the AUC of the live vaccine virus shedding determined by 50% tissue culture infectious dose (TCID ) on MDCK cells at 33 degrees C | nasal swab at 4 days post vaccination
The primary endpoint for assessment of the live attenuated vaccine take will be the AUC of the live vaccine virus shedding determined by 50% tissue culture infectious dose (TCID ) on MDCK cells at 33 degrees C | nasal swab obtained at 7 days post vaccination

SECONDARY OUTCOMES:
The AUC of nasopharyngeal shedding assessed by quantitative rtRT-PCR | swabs will be obtained on day 2 post vaccination
The frequency and magnitude of serum hemagglutination-inhibition (HAI), ELISA, and neutralizing antibody response to vaccine | at day 28
The frequency and magnitude of hemagglutinin-specific mucosal IgA response assessed by ELISA on nasal secretions | day 28
The frequency and magnitude of antibody secreting cell and memory B cells developing after vaccination | on day 7
Development of specific local and systemic symptoms occuring after vaccine | for 7 days post each vaccination
The AUC of nasopharyngeal shedding assessed by quantitative rtRT-PCR | swab obtained at day 4 post vaccination
The AUC of nasopharyngeal shedding assessed by quantitative rtRT-PCR | swab obtained at day 7 post vaccination
The frequency and magnitude of serum hemagglutination-inhibition (HAI), ELISA, and neutralizing antibody response to vaccine | at day 56
The frequency and magnitude of hemagglutinin-specific mucosal IgA response assessed by ELISA on nasal secretions | at day 56
The frequency and magnitude of antibody secreting cell and memory B cells developing after vaccination | on day 35

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Vaccine Research Unit Room 3-5000, Rochester, New York, United States

REFERENCES:
- [Background] Hancock K, Veguilla V, Lu X, Zhong W, Butler EN, Sun H, Liu F, Dong L, DeVos JR, Gargiullo PM, Brammer TL, Cox NJ, Tumpey TM, Katz JM. Cross-reactive antibody responses to the 2009 pandemic H1N1 influenza virus. N Engl J Med. 2009 Nov 12;361(20):1945-52. doi: 10.1056/NEJMoa0906453. Epub 2009 Sep 10. PMID 19745214
- [Background] Shinde V, Bridges CB, Uyeki TM, Shu B, Balish A, Xu X, Lindstrom S, Gubareva LV, Deyde V, Garten RJ, Harris M, Gerber S, Vagasky S, Smith F, Pascoe N, Martin K, Dufficy D, Ritger K, Conover C, Quinlisk P, Klimov A, Bresee JS, Finelli L. Triple-reassortant swine influenza A (H1) in humans in the United States, 2005-2009. N Engl J Med. 2009 Jun 18;360(25):2616-25. doi: 10.1056/NEJMoa0903812. Epub 2009 May 7. PMID 19423871
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Belshe RB, Edwards KM, Vesikari T, Black SV, Walker RE, Hultquist M, Kemble G, Connor EM; CAIV-T Comparative Efficacy Study Group. Live attenuated versus inactivated influenza vaccine in infants and young children. N Engl J Med. 2007 Feb 15;356(7):685-96. doi: 10.1056/NEJMoa065368. PMID 17301299
- [Background] Maassab HF. Biologic and immunologic characteristics of cold-adapted influenza virus. J Immunol. 1969 Mar;102(3):728-32. No abstract available. PMID 5773321
- [Background] Chanock RM, Murphy BR. Use of temperature-sensitive and cold-adapted mutant viruses in immunoprophylaxis of acute respiratory tract disease. Rev Infect Dis. 1980 May-Jun;2(3):421-32. doi: 10.1093/clinids/2.3.421. PMID 6997969
- [Background] Boyce TG, Gruber WC, Coleman-Dockery SD, Sannella EC, Reed GW, Wolff M, Wright PF. Mucosal immune response to trivalent live attenuated intranasal influenza vaccine in children. Vaccine. 1999 Aug 20;18(1-2):82-8. doi: 10.1016/s0264-410x(99)00183-8. PMID 10501238
- [Background] Sasaki S, Jaimes MC, Holmes TH, Dekker CL, Mahmood K, Kemble GW, Arvin AM, Greenberg HB. Comparison of the influenza virus-specific effector and memory B-cell responses to immunization of children and adults with live attenuated or inactivated influenza virus vaccines. J Virol. 2007 Jan;81(1):215-28. doi: 10.1128/JVI.01957-06. Epub 2006 Oct 18. PMID 17050593
- [Background] Cox RJ, Brokstad KA, Zuckerman MA, Wood JM, Haaheim LR, Oxford JS. An early humoral immune response in peripheral blood following parenteral inactivated influenza vaccination. Vaccine. 1994 Aug;12(11):993-9. doi: 10.1016/0264-410x(94)90334-4. PMID 7975853
- [Background] He XS, Holmes TH, Zhang C, Mahmood K, Kemble GW, Lewis DB, Dekker CL, Greenberg HB, Arvin AM. Cellular immune responses in children and adults receiving inactivated or live attenuated influenza vaccines. J Virol. 2006 Dec;80(23):11756-66. doi: 10.1128/JVI.01460-06. Epub 2006 Sep 13. PMID 16971435